CLINICAL TRIAL: NCT00974467
Title: Evaluating a Website for Parents of Injured Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008-4-5932
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2012-01

CONDITIONS: Acute Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- After The Injury website (Experimental)
  Interventions: Behavioral: After The Injury website
- Usual care (Other): Treatment as usual
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: After The Injury website — Parents participate in a web-based prevention intervention, which provides education and tips specific to coping with a child's injury.
  Arms: After The Injury website
Other: Control — Usual hospital care provided.
  Arms: Usual care

SUMMARY:
The purpose of the current protocol is to evaluate the ability of the AfterTheInjury website to increase parent knowledge and skills.

DETAILED DESCRIPTION:
The purpose of the current protocol is to evaluate the ability of the AfterTheInjury website to increase parent knowledge and skills. Primary objective is to compare website condition vs control with regard to (a) immediate parent learning outcomes and (b) coping assistance provided by parents as reported at 6 wks. Secondary objective is to compare conditions as above with regard to child and parent PTS symptoms at 6 wks.

ELIGIBILITY:
Inclusion Criteria:

1. Children age 6 through 17 who sustained an injury within the past 2 months and their parents.
2. Have access to the Internet at home (for Stage 3 only)

Exclusion Criteria:

1. Parent does not read or understand English
2. Child's injury is due to participation in organized sports
3. Child's injury is due to suspected abuse or family violence

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Scores on measure of parent knowledge re: traumatic stress and coping assistance. | 6 wks post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Kassam-Adams, Ph.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States